CLINICAL TRIAL: NCT03923504
Title: Improving Exercise Capacity With a Tailored Physical Activity Intervention in Lymphoma and Breast Cancer Patients Undergoing Treatment
Brief Title: Improving Exercise Capacity With Tailored Physical Activity in Lymphoma & Breast Cancer Patients Undergoing Tx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCC-19-14621
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Hodgkin Lymphoma; Non-hodgkin Lymphoma; Lymphoma; Breast Cancer
Keywords: Physical Activity Intervention; Healthy Living Intervention; Health-related Quality of Life
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (PAI) (Active Comparator): Tailored multi-level physical activity intervention (PAI) on exercise capacity, cardiovascular and cognitive function, health-related quality of life (QOL), strength and fatigue among lymphoma and breast cancer patients undergoing active treatment with anthracycline based chemotherapy (anthra-bC).
  Interventions: Other: Physical Activity Intervention (PAI)
- Healthy Living Control Group (Active Comparator): Healthy living intervention (HLI) on exercise capacity, cardiovascular and cognitive function, health-related quality of life (QOL), strength and fatigue among lymphoma and breast cancer patients undergoing active treatment with anthracycline based chemotherapy (anthra-bC).
  Interventions: Other: Healthy Living Control

INTERVENTIONS:
Other: Physical Activity Intervention (PAI) — Those who opt-in to attend in-person study visits and to undergo COVID testing will also complete an MRI exam and CPET testing. Participants unwilling to have COVID testing done will only complete an MRI exam and home-based testing. All testing will take place either within 6 weeks of initiating systemic treatments or within 8 weeks of completing radiation then at 3 & 6 months. Patients may participate in 1-2 training sessions per week offered under the direct supervision of a master's level clinical exercise physiologist, as well as 1-2 sessions at home. PAI sessions consist of slow aerobic warm-up, followed by 20 minutes of strength training,15 minutes of progressive intensity aerobic exercise (AE), and then 10 minutes of stretching for cool-down. Participants will have the ability to participate in training sessions facilitated via online channels at home.
  Arms: Physical Activity Intervention (PAI)
Other: Healthy Living Control — Patients randomized to the control arm will either attend online sessions via secure video conferencing (e.g. Zoom) or telephone or to come to a centralized meeting location (if safety allows) to participate in organized health workshops. Session attendance will be required 2 times/month (over the 6 months). Make up sessions will be offered for those participants who have to miss a group session. Each session lasts 60 minutes and matches the number of visits made by the PAI group as much as possible.
  Arms: Healthy Living Control Group

SUMMARY:
To provide critical participant enrollment data necessary to complete a larger definitive clinical trial in the future.

DETAILED DESCRIPTION:
This study is a 2-arm, parallel design, single-blind randomized controlled pilot study designed to compare the effects of a tailored multi-level physical activity intervention (PAI) vs healthy living intervention (HLI) on exercise capacity, cardiovascular and cognitive function, health-related quality of life (QOL), strength and fatigue among lymphoma and breast cancer patients undergoing active treatment with anthracycline based chemotherapy (anthra-bC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18-85 years old
* Stage I-IV Hodgkin's (HL) or Non-Hodgkin's Lymphoma (NHL) or I-III Breast Cancer patients who are receiving (within 6 weeks of initiation) or are scheduled to receive potentially cardiotoxic systemic therapies (e.g. chemotherapy regimens [anthracyclines, trastuzumab]), immuno-therapies (immune checkpoint inhibitors [ICI's]), hormonal therapies (aromatase inhibitors) or radiation (within 8 weeks of completion).

Exclusion Criteria:

* Evidence of COVID19 within the last 60 days or recent (21 days) exposure to close personal contact who has tested positive for COVID19.
* Uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg)
* A recent history of alcohol or drug abuse
* Inflammatory conditions such as lupus or inflammatory bowel disease, or another medical condition that might compromise safety or successful completion
* Other exclusions include those with contraindications to MRI; unstable angina; inability to exercise on a treadmill or stationary cycle; significant ventricular arrhythmias (>20 PVCs/min due to gating difficulty); atrial fibrillation with uncontrolled ventricular response; acute myocardial infarction within 28 days; claustrophobia; pregnancy; those unable to provide informed consent (able to read and write English); or moving within 12 mos. of enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Assessment of Patient Interest in Protocol | 6 Months
  Feasibility for a larger study will be determined by the number of patients that agree to participate in the trial.
Assessment of Patient Compliance | 6 Months
  Data collected will determine how many patients complete all protocol activities to determine feasibility of the interventions.
Assessment of Patient Response to Interventions | 6 Months
  Examination of qualitative data to evaluate positive and negative influences on adherence and to refine the intervention for a future large scale utilizing recorded interviews with each of the accrued subjects.

SECONDARY OUTCOMES:
Assessment of Cardiac Output | 6 Months
  Assessment of the subject's peak exercise cardiac output at the initial visit, then at 3 and 6 months after starting Anthracycline-based Chemotherapy (Anth-bC) utilizing Magnetic Resonance Imaging (MRI) variables, and Cardiopulmonary Exercise Testing (CPET).
Assessment of Oxygen Output | 6 Months
  Assessment of oxygen output will be determined by using measurements from maximal oxygen intake, and a six-minute walk test to obtain exercise capacity.
Assessment of Health Related Quality of Life | 6 Months
  Health related quality of life will be measured using the Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) questionnaire to assess disease-specific health related quality of life (HRQoL). The FACT-Lym scale measures HRQoL using a forty-two question assessment that measures physical well-being, social well-being, and emotional well-being. Each item on the FACT-Lym scale is scored from 0 (Not at all) to 4 (very much). All items are summed to create a total score (range 0-108) and sub-scales may be scored separately for questions related to physical well-being (range 0-28), social well-being (range 0-28), emotional well-being (range 0-24), functional well-being (range 0-28), and for lymphoma specific additional concerns (range 0-60). Negatively worded items are reverse scored prior to summing so that higher sub-scale and total scores indicate better QoL.
Assessment of Fatigue | 6 Months
  Fatigue will be assessed by utilizing the Functional Assessment of Cancer Therapy-Fatigue scale (FACT-fatigue) assess fatigue. The FACT-fatigue scale assesses cancer related fatigue using a thirteen question scale. Each item on the FACT-Fatigue scale is scored from 0 (not at all) to 4 (very much). All items on the scale are summed to provide a total score for fatigue (range 0-52)
Assessment of General Health | 6 Months
  The MOS 36-item Short Form Health Survey (SF-36) will also be used to to measure subject's general health. All items on the SF-36 are scored from 1 (excellent) to 5 (poor). Scores are calculated for eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  All items are scored so that a high score defines a more favorable health state. each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Assessment for Anemia | 6 Months
  Blood will be obtained at each study visit to assess hemoglobin and hematocrit levels.
Assessment of Renal Function | 6 Months
  Blood will be obtained at each study visit to assess for renal (kidney) dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lucas, Ph.D., Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Virginia Commonwealth University Community Memorial Health Center, South Hill, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NCT01719562: MRI in Detecting Heart Damage in Patients With Cancer Receiving Chemotherapy With Exercise Capacity Addendum — https://clinicaltrials.gov/ct2/show/NCT01719562?term=NCT01719562&draw=2&rank=1

DOCUMENTS (1):
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03923504/ICF_000.pdf